CLINICAL TRIAL: NCT01083862
Title: Impact of Health Literacy on Outcomes and Effectiveness of Shared Decision Making Programs in Patients With Chronic Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Foundation for Informed Medical Decision Making (Other)
Responsible Party: Principal Investigator, Mark Eckman, M.D., Professor Emeritus, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FIMDM-CS09052/GR090501
Record Dates: First submitted 2010-03-05; First posted 2010-03-10 (Estimated); Last update posted 2023-12-07 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease
Keywords: Health literacy; patient education; health behaviors; chronic disease management; shared decision-making; patient-centered decision making
MeSH Terms: conditions — Coronary Artery Disease; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational Intervention - Video & Text (Experimental): Educational Intervention - Video & Text describing "Living with Coronary Artery Disease."
  Interventions: Behavioral: Educational Intervention - Text plus DVD/VHS
- Educational Intervention - Text Only (Active Comparator): Educational Intervention - Text Only describing "Living with Coronary Artery Disease."
  Interventions: Behavioral: Educational Intervention - Text Only

INTERVENTIONS:
Behavioral: Educational Intervention - Text plus DVD/VHS — In conjunction with a scheduled clinical visit, consenting patients spent roughly 40 minutes viewing a video program developed by the Foundation for Informed Decision Making (FIMDM), describing life-style and behavior modification for patients "Living with Coronary Artery Disease." They also were given a booklet on the same subject material written at a 5th grade level.
  Arms: Educational Intervention - Video & Text
Behavioral: Educational Intervention - Text Only — In conjunction with a scheduled clinical visit, consenting patients spent roughly 40 minutes reading a booklet developed by the Foundation for Informed Decision Making (FIMDM), describing life-style and behavior modification for patients "Living with Coronary Artery Disease." Subject material was written at a 5th grade level.
  Arms: Educational Intervention - Text Only

SUMMARY:
Study objective was to explore the impact of health literacy on effectiveness of an educational intervention describing life-style and behavior modification for patients "Living with Coronary Artery Disease." Our hypothesis was that a VHS/DVD version of this educational program would be "superior" to printed material alone in its impact on patients' knowledge about coronary artery disease and important life-style changes. Furthermore, we believed this effect would be most notable among patients with low health literacy. We also were interested in the impact of the interventions on secondary outcomes including - health behaviors, health outcomes and patients' subjective experiences.

DETAILED DESCRIPTION:
187 patients with coronary artery disease (CAD) were randomized to one of two educational interventions prior to scheduled ambulatory visit: VHS/DVD plus printed booklet; or booklet alone. Main measures included health literacy, CAD knowledge assessment; clinical outcomes and health behaviors including - blood pressure, weight, smoking status, exercise and dietary habits.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18,
* Diagnosis of ischemic heart disease.

Exclusion Criteria:

* Nursing home resident,
* Did not speak English, or
* Had a significant visual impairment that precluded their ability to read or watch television.

Ages: 18 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2005-10; Primary Completion 2007-10 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
cardiovascular disease knowledge assessment score | immediate and 6 months
  knowledge assessment performed prior to educational intervention, immediately after educational intervention and clinician visit, and once more at approximately 6 months

SECONDARY OUTCOMES:
Smoking status | over 6 months of study
  Noted initial smoking status and followed whether patients continued to smoke and if so, how much
Diet | Over six months of study
  Performed MEDFICTs dietary assessment at study start and at study completion, roughly 6 months later
Exercise | Over 6 months of study
  Performed PASE exercise survey at study start and at study completion.
Weight | over 6 month study
  Measured weight at study start and at study completion
Blood Pressure | over 6 months of study
  Measured blood pressure at study start and at study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Eckman, MD, Principal Investigator — University of Cincinnati
Locations (1):
- General Internal Medicine Hoxworth Practices, Cincinnati, Ohio, United States